CLINICAL TRIAL: NCT01965795
Title: Effects of Whole Coffee Fruit Concentrate On Cognition and Mood In Healthy Adults: A Pilot Clinical Study
Brief Title: Whole Coffee Fruit Concentrate Pilot Study 1
Acronym: WCFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Applied BioClinical Inc. (Industry)
Responsible Party: Principal Investigator, Edythe London, Ph.D., University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-001426
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Brain-derived Neurotrophic Factor (BDNF); Cognitive Function; Affect
Keywords: Brain-derived neurotrophic factor; Cognitive function; Dietary supplement; Coffee plant extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrim (Placebo Comparator): Nutrim will be capsulated in size 1 gelatin capsules, white and blue, distributed in brown plastic bottles (28 caps/bottle: enough for 14 days of treatment). The first bottle will be provided at the time of randomization, and the second bottle will be provided on day 14 for dosing on days 15-28. The bottle will be labeled with the ABC logo and treatment code.
  A dose of 100 mg will be administered twice daily (once before breakfast and again before dinner).
  Interventions: Dietary Supplement: Nutrim
- Whole Coffee Fruit Concentrate (WCFC) (Experimental): WCFC is in powder form, and will be capsulated in size 1 gelatin capsules, white and blue, distributed in brown plastic bottles (28 caps/bottle: enough for 14 days of treatment). The first bottle will be provided at the time of randomization, and the second bottle will be provided on day 14 for dosing on days 15-28. The bottles will be labeled with the ABC logo and treatment code.
  A dose of 100 mg will be administered twice daily (once before breakfast and again before dinner).
  Interventions: Dietary Supplement: Whole Coffee Fruit Concentrate (WCFC)

INTERVENTIONS:
Dietary Supplement: Whole Coffee Fruit Concentrate (WCFC) — Neurfactor is a powder dietary supplement patented by Futureceuticals, in which the active ingredient is WCFC. It is hypothesized that the whole fruit of the coffee plant, Coffea arabica, has very unique, important benefits for healthy aging not available from regular coffee, other coffee extracts, green coffee bean extracts, caffeine, or other leading botanicals. NeuroFactor is thought to increase Brain-Derived Neurotrophic Factor, a protein vital for neuron development, repair and protection and essential for learning, memory, alertness, controlling body weight, and energy metabolism.
  Other Names: NeuroFactor
  Arms: Whole Coffee Fruit Concentrate (WCFC)
Dietary Supplement: Nutrim — Nutrim is an oat bran powder Nutrim is hypothesized to bestow a number of benefits such as cardiovascular health, glucose management and healthy digestion. However, improved cognition is not one of the hypothesized benefits. This product is free of caffeine and stimulants.
  Arms: Nutrim

SUMMARY:
The purpose of this pilot study is to evaluate the potential effects of whole coffee fruit concentrate (WCFC, Neurofactor), a product that elevates circulating brain-derived neurotrophic factor (BDNF), on cognition and mood in healthy adults.

The projected outcome of this study is that self-administration of Neurofactor for 28 days (or even 14 days) will be associated with an improvement in mood and scores on cognitive tests, and that the change will exceed that observed with administration of Nutrim (placebo).

Volunteers will be recruited from the greater Los Angeles community. Participants will be middle-aged nonsmokers, in good health, and between the ages of 40-55 to enhance the chance of demonstrating pro-cognitive effects. Younger participants, whose cognitive performance is expected to be higher, may perform at a ceiling level, with less room for improvement by the product under study.

Participants who call our lab will be told about the study in more detail, and will complete a 5 minute phone screener to determine preliminary eligibility. After the initial telephone screening, participants will visit Dr. London's laboratory at UCLA to provide written informed consent.

The first study visit will be an in-person screening visit to determine full eligibility. The evaluation will include a psychiatric diagnostic interview, using the SCID, blood tests, urine samples (to test for drug use and pregnancy). Participants will also be interviewed about their prior and current drug use, including tobacco use. In addition, participants will be interviewed about the nature of their employment and physical exercise habits: endurance training has been shown to increase plasma BDNF in young men.

Participants meeting the inclusion criteria will attend the Semel Institute for Neuroscience and Human Behavior at UCLA to take part in baseline measurements, and to be randomized to receive either WCFC or placebo. During the active treatment time (28 days), they will visit the UCLA Semel Institute on a weekly basis. At each of these weekly visits, questionnaires regarding compliance will be completed, and blood samples will be taken for assay of BDNF. A cognitive test battery and mood-rating scales will be completed at baseline and at 14 and 28 days of treatment. At the midpoint assessment (14 days) and at completion of treatment (28 days) blood will be drawn for assay of a blood chemistry panel (as at baseline) as well as for biomarkers in addition to BDNF.

DETAILED DESCRIPTION:
Participants (n=23; 20 completing with usable data) will come to UCLA for 1 in-person screening visit and 4 weekly study visits, culminating in a total of 5 study visits. Those who meet eligibility criteria will take part in a baseline test session (before randomization) to collect cognitive and behavioral data as well as baseline plasma BDNF level. There will also be two test sessions at 14 and 28 days of treatment to collect data on the effects of the active and placebo treatments. The questionnaires, cognitive tasks, and diagnostic interviews will be conducted on an outpatient basis at the Semel Institute for Neuroscience and Human Behavior, and the medical procedures will take place at the UCLA Clinical and Translational Research Center (CTRC).

In-person screening procedures:

First, investigators will thoroughly explain the study and obtain informed consent from interested participants. Immediately after consent is obtained, the following questionnaires/ diagnostic interviews will be completed:

* Study Admission & Intake Form- This questionnaire administered at intake collects demographic information (i.e. ethnicity, education, employment), general and mental health history, as well as substance abuse history. This questionnaire takes approximately 15-45 min to complete.
* Psychiatric evaluation using the SCID-IR-TR. The SCID will be administered during intake screening to determine whether the participant meets the DSM-IV-TR criteria for drug dependence and to rule out any major psychiatric disorders (e.g., affective disorders, schizophrenia; Spitzer et al., 1995).
* The International Physical Activity Questionnaires (IPAQ). The purpose of the IPAQ (Craig et al., 2003) is to record any exercise that participants engage in as this may impact findings. It takes approximately 5 min to complete.

Urine testing (40 ml) will be done to test for pregnancy (females only) and drugs of abuse. Urine testing will be done at screening as well as each of the study visits. Once the urine has been analyzed, it will be disposed of in a sanitary manner.

Medical Procedures completed during in-person screening:

Participants will give a blood sample taken for Rapid Plasma Reagin (RPR), and Hepatitis B and C testing [25-ml sample to including a complete chemistry panel (5 ml), hepatic panel (3 ml), Hepatitis B and C, RPR test (7 ml), plasma BDNF (0.1 ml)]. The study physician will inform participants of the implications if their status for RPR, hepatitis B or hepatitis C test results is positive, and will refer participants to further information. Study staff will inform participants with negative RPR, hepatitis B and hepatitis C test results of their health status. Height and weight will be assessed, as body mass index (BMI) values provide inclusion criteria (18 ≤ BMI ≥ 25 kg/m2). In addition, vital signs such as heart-rate (ECG), pulse, and blood pressure will be measured. Plasma BDNF (and other biomarkers) will be measured by a blood sample (finger stick) obtained prior to, and at each weekly visit to UCLA after initiating WCFC or placebo administration.

The maximum time period allowable between the screening visits and attendance at the UCLA CTRC will be 4 weeks. If this time elapses, the potential subject will be screened again.

Study Visit Timeline:

Day Up to -28: Telephone screening Day 0- In-person medical screening, baseline cognitive testing session and rating of subjective mood states. BDNF assay. Randomization to group, and initiation of WCFC/placebo treatment, with 14-day supply provided to the participant.

Day 7- Collection of compliance questionnaire, BDNF assay. Day 14- Cognitive testing and rating of subjective mood states. Collection of compliance questionnaire; re-supply WCFC/placebo; and phlebotomy for blood chemistry and assay of BDNF and other biomarkers.

Day 21- Collection of compliance questionnaire, BDNF assay. Day 28- Completion of WCFC/placebo treatment. Final cognitive testing session and rating of subjective mood states. Collection of compliance questionnaire. Phlebotomy for blood chemistry, and assay of BDNF and other biomarkers.

Study Visit Procedures (~2-3 hrs):

Participants meeting the inclusion criteria will be randomized to receive either WCFC or placebo. During the active treatment time (28 days), they will visit the UCLA Semel Institute on a weekly basis. On day 0 (at baseline) and day 14, WCFC or placebo will be provided, in amounts sufficient for a 2-week supply, so that they can self-administer the respective treatments. At each of these weekly visits, questionnaires regarding compliance will be completed, and blood samples will be taken for assay of BDNF. A cognitive test battery and mood-rating scales will be completed at baseline and at 14 and 28 days of treatment. At the midpoint assessment (14 days) and at completion of treatment (28 days) blood will be drawn for assay of a blood chemistry panel (as at baseline) as well as for biomarkers in addition to BDNF.

Nutraceutical Administration and Dose Justification:

WCFC (NeurofactorTM): A dose of 100 mg will be administered twice daily (once before breakfast and again before dinner). The dose was chosen on the basis of published work from Applied Bioclinical, Inc. (Reyes-Izquierdo et al., 2013; Pietrzkowski et al., in press). Specifically, Reyes-Izquierdo and colleagues (2013) reported that 100 mg of WCFC resulted in increased plasma BDNF by 143% from baseline (n=10, healthy adults aged between 18 and 55 years old). More recently Pietrzkowski and co-workers (unpublished manuscript in press) observed a 90% increase in plasma BDNF during the first 60 minutes after a single 100 mg dose of WCFC. The effect is sustained for 2-3 hours. Therefore, testing will always take place in the morning within 2 hours of WCFC ingestion with breakfast. As a quality control measure, WCFC batches will be tested to delineate the same chemical profile of polyphenols to make sure that if more than one batch is used, the chemical profiles are identical between batches.

Placebo: The placebo will be Nutrim®, supplied by Abclinical and administered twice daily, identical to WCFC treatment (other participant group).

Both WCFC and placebo are in powder form, and will be capsulated in size 1 gelatin capsules, white and blue, distributed in brown plastic bottles (28 caps/bottle: enough for 14 days of treatment). The first bottle will be provided at the time of randomization, and the second bottle will be provided on day 14 for dosing on days 15-28. The bottles will be labeled with the ABC logo and treatment code ABC#7UCLA01 and ABC#7UCLA12.

The following questionnaires that assess mood will be administered during each of the study sessions:

* HAM-D- The Hamilton Depression Rating Scale is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Assessment time is estimated at 20 minutes. The HAM-D has been used previously, showing a correlation between increased plasma BDNF and improved (decreased) HAM-D scores (e.g., Shimizu et al., 2003, Gonul et al., 2005, Aydemir et al., 2005, Yoshimura et al., 2007).
* PANAS- The Positive and Negative Affect Schedule (Watson et al., 1988) is a 20-item questionnaire that comprises two mood scales, one measuring positive affect and the other measuring negative affect. Each item is rated on a 5-point scale ranging from 1 = very slightly or not at all to 5 = extremely to indicate the extent to which the respondent has felt this way in the indicated time frame. The participant will be instructed to provide these ratings of his or her affective state at the time of assessment.
* Adverse Events Log- At each visit after randomization, any adverse events that occur will be recorded, and evaluated in terms of frequency and severity (mild, moderate, severe) using this form.

The following cognitive tests will be administered during each of the study sessions:

* Hopkins Verbal Learning Test- Revised (HVLT-R): This task is an assessment of verbal memory.
* Continuous Performance Test (CPT): This computer task is an assessment of attention & inhibition.
* Spatial Sternberg: This computer task is an assessment of spatial short term memory.
* Letter Number Sequencing: This task in an assessment of working memory.
* Attention Networks Task: This computer task is an assessment of attention & inhibition.
* Verbal fluency: This task is an assessment of executive function.
* Finger Tapping: This task is an assessment of psychomotor speed.

These tests will assess multiple cognitive domains, and the total battery of tests will take approximately 1.5 hours to complete. Thus, the burden on participants will be low. Participants will be trained on the tasks before the baseline measurement is taken to reduce the effects of learning on performance.

Biochemical Measures:

The biochemical measurements that will be performed during the study will be the determination of plasma BDNF at baseline (conducted during medical screening procedure) and at each weekly visit following the initiation of WCFC and placebo administration, and assay of other biomarkers in serum at the 14- and 28-day test points. Determination of plasma BDNF must be performed at the same time of day for all subjects at all time-points, due to diurnal variation in plasma BDNF levels (Piccini et al., 2008). Weekly BDNF data will be used as an index of compliance with WCFC administration. Data at baseline, 14 days and 28 days will be used in tests of association with behavioral measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be 45-55 years old. Investigators have selected an age range of 40-55 years to enhance the chance of demonstrating pro-cognitive effects. Younger participants, whose cognitive performance is expected to be higher, may perform at a ceiling level, with less room for improvement by the product under study. An emerging body of data suggests speculation that natural polyphenols can combat age-related cognitive decline, which is often accompanied by depression and potentially by reduced levels of hippocampal neurogenesis (Ogle et al., 2013).
* Language: Subjects must be fluent in English (in order to provide consent, complete questionnaires,& cognitive testing)
* BMI: Body mass index values ≥ 18 kg/m2 and ≤ 25 kg/m2
* Vital signs: must be within the clinically acceptable normal range (i.e., resting pulse between 50 and 90 beats/min (bpm), blood pressures between 85-150 mm Hg systolic and 45-90 mm Hg diastolic
* Pregnancy prevention: if female, must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal,) or agree to use a reliable form of contraception (e.g., birth control pills, intrauterine device, condoms, or spermicide) during the trial and to provide a negative pregnancy urine test before randomization.

Exclusion Criteria:

* Certain medical conditions: Participants may not have a medical condition that, in the study physician's judgment, may interfere with safe participation (e.g., active tuberculosis, unstable cardiac, renal, pulmonary or liver disease, unstable diabetes)
* Neurological disorder: Participants should not have a current neurological disorder (e.g., organic brain disease, dementia) or a medical history which would make compliance difficult or would compromise informed consent
* Psychiatric disorder: must not have an Axis I psychiatric disorder as assessed by the Structured Clinical Inventory for DSM-IV-TR (SCID)
* Suicide Attempt(s): Participants may not have a history of attempted suicide in the past 3 years and/or serious suicidal intention or plan in the past month as assessed by the SCID
* Prescription medications: must not be taking a prescription medication that can affect brain function
* Alcohol dependence: Must not have a history of alcohol dependence within the past 3 years
* Pregnancy or nursing
* Heart abnormality: Participants should not have a clinically significant heart disease or hypertension; ECG showing cardiac ischemia or other clinically significant abnormality
* Smoking: Participants must be current non-smokers
* Illicit drug use: Participants must not have a current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV-TR
* Other: Participants may not have any other circumstance that, in the opinion of investigators, would compromise safety

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Biochemical measures of brain-derived neurotrophic factor (BDNF) | 28 days
  One of the outcome measures will be the determination of plasma BDNF at 3 different time points within a 28 day period via a blood sample.

SECONDARY OUTCOMES:
Cognitive Functioning | 28 days
  Tests of cognitive function will be given on day 0, 14, and 28.
  Tests include:
  * Hopkins Verbal Learning Test- Revised (HVLT-R): assessment of verbal memory.
  * Continuous Performance Test (CPT): assessment of attention & inhibition.
  * Spatial Sternberg: assessment of spatial short term memory.
  * Letter Number Sequencing: assessment of working memory.
  * Attention Networks Task: assessment of attention & inhibition.
  * Verbal fluency: assessment of executive function.
  * Finger Tapping: assessment of psychomotor speed.

OTHER OUTCOMES:
Affect | 28 days
  The following mood assessments will be given on days 0, 14, & 28:
  * HAM-D. The Hamilton Depression Rating Scale is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Assessment time is estimated at 20 minutes.
  * PANAS. The Positive and Negative Affect Schedule (Watson et al., 1988) is a 20-item questionnaire that comprises two mood scales, one measuring positive affect and the other measuring negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, PhD, Principal Investigator — Professor in Residence
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Reyes-Izquierdo T, Nemzer B, Shu C, Huynh L, Argumedo R, Keller R, Pietrzkowski Z. Modulatory effect of coffee fruit extract on plasma levels of brain-derived neurotrophic factor in healthy subjects. Br J Nutr. 2013 Aug 28;110(3):420-5. doi: 10.1017/S0007114512005338. Epub 2013 Jan 14. PMID 23312069
- [Background] Yoshimura R, Mitoma M, Sugita A, Hori H, Okamoto T, Umene W, Ueda N, Nakamura J. Effects of paroxetine or milnacipran on serum brain-derived neurotrophic factor in depressed patients. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jun 30;31(5):1034-7. doi: 10.1016/j.pnpbp.2007.03.001. Epub 2007 Mar 7. PMID 17459550
- [Background] Gonul AS, Akdeniz F, Taneli F, Donat O, Eker C, Vahip S. Effect of treatment on serum brain-derived neurotrophic factor levels in depressed patients. Eur Arch Psychiatry Clin Neurosci. 2005 Dec;255(6):381-6. doi: 10.1007/s00406-005-0578-6. Epub 2005 Apr 6. PMID 15809771
- [Background] Shimizu E, Hashimoto K, Okamura N, Koike K, Komatsu N, Kumakiri C, Nakazato M, Watanabe H, Shinoda N, Okada S, Iyo M. Alterations of serum levels of brain-derived neurotrophic factor (BDNF) in depressed patients with or without antidepressants. Biol Psychiatry. 2003 Jul 1;54(1):70-5. doi: 10.1016/s0006-3223(03)00181-1. PMID 12842310
- [Background] Piccinni A, Marazziti D, Catena M, Domenici L, Del Debbio A, Bianchi C, Mannari C, Martini C, Da Pozzo E, Schiavi E, Mariotti A, Roncaglia I, Palla A, Consoli G, Giovannini L, Massimetti G, Dell'Osso L. Plasma and serum brain-derived neurotrophic factor (BDNF) in depressed patients during 1 year of antidepressant treatments. J Affect Disord. 2008 Jan;105(1-3):279-83. doi: 10.1016/j.jad.2007.05.005. Epub 2007 Jun 5. PMID 17553570
- [Background] Ogle WO, Speisman RB, Ormerod BK. Potential of treating age-related depression and cognitive decline with nutraceutical approaches: a mini-review. Gerontology. 2013;59(1):23-31. doi: 10.1159/000342208. Epub 2012 Aug 30. PMID 22947921